CLINICAL TRIAL: NCT04111198
Title: Epicardial Fat Tissue and Severity of Coronary Artery Disease in Diabetic vs Non Diabetic Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bakeer Mohamed Bakeer (Other)
Responsible Party: Sponsor-Investigator, Bakeer Mohamed Bakeer, Resident, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Epicardial fat tissue
Record Dates: First submitted 2019-09-29; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Epicardial Fat Tissue
Keywords: Epicardial fat tissue; Cardiac MRI; Coronary Artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- coronary artery disease in diabetic and non diabetic patients
  Interventions: Radiation: Cardiac MRI

INTERVENTIONS:
Radiation: Cardiac MRI — Cardiac MRI

SUMMARY:
correlation between EFT volume measured by Cardiac MRI and the angiographic severity of coronary artery disease (Syntax Score) in diabetic vs non diabetic CAD population and detect if there is a cut off value for each group that could predict higher risk.

DETAILED DESCRIPTION:
Epicardial fat tissue (EFT) is is most commonly defined as adipose tissue surrounding the heart, located between the myocardium and the visceral layer of pericardium Once considered only as a mere storage compartment, the adipose tissue is now recognized for its extensive metabolic and endocrine function, EFT is a storage fat that covers 80% of the heart's surface, representing 20% of the organ total weight, EFT is considered to be a part of visceral adipose tissue. This fat is a major source of biomolecules and compartmentalized production of cytokines and hormones, acting as a localized gland.

Moreover, EFT and the underlying myocardium share the same microcirculation, suggesting a close and strong interaction between these two structures, it regulates heart and blood vessel physiologically, via paracrine and vasocrine mechanisms. It has also been reported that EFT acts as important energy reservoir for cardiomyocytes, which depend on fatty acids oxidations as energy source especially during periods of high demand.

Although EFT is needed for heart muscle function, in recent decades it has been published that increased thickness greatly enhances the risk of developing CVD and metabolic syndrome, becoming a new pharmacological target for primary and secondary prevention strategies. Therefore, the measurement of epicardial fat deposition is important. In terms of modulation, the use of statins could function as a possible treatment to help decrease the volume of EFT beside stabilization of atherosclerotic plaques.

Detection and quantification of EFT require a variety of useful imaging techniques, including 2-dimensional (2D) echocardiography, non-contrast computed tomography (CT) and magnetic resonance imaging (MRI) . Since fat tissue generates a strong MRI signal, both thickness and volume of epicardial fat can be easily measured with this modality.

Clinical research found that it was related to coronary artery disease, where it was found to be independently and linearly associated with CAD and its severity, atrial fibrillation as well as myocardial dysfunction.

It is known that abnormally accumulated visceral fat is a risk factor for insulin resistance, which can reduce insulin sensitivity, increase the expression and secretion of proinflammatory cytokines in adipose tissue and promote the development of DM and cardiovascular diseases. Since EFT is a part of the visceral fat, it carries that risk.

Regarding relation to CAD in DM, there have been conflicting data.

Maniam et al reported that EFT was higher in non-diabetics with CVD, but not in T2DM with or without CVD. This suggests EFT may play a greater role in CVD in non-diabetics than those with T2DM.

However, in the past few years, several other studies have reported that EFT is abnormally increased in DM patients. However, small sample sizes and potential confounders (such as differences in EFT measurements and DM typing) were thought to affect the strength of previous evidence.

A metanalysis conducted suggests that the amount of EFT is significantly higher in DM patients than in non-DM patients.

Another study addressing mainly type 1 DM found that Long-term survivors of T1DM have a higher prevalence of coronary atherosclerosis compared to controls but EFT volume was not associated with coronary atherosclerosis in T1DM patients.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Patients presenting for cardiac MRI unit in Assiut University Hospital for viability assessment.
* Having diagnostic coronary angiography done or to be done within a 3 months of the cardiac MRI study

Exclusion Criteria:

* patients not having CA within the aforementioned time limits. Other classical contraindications of cardiac MRI including: MRI non-conditional devices, claustrophobia and eGFR> 30 ml/sec/1.73 m2 BSA. (NB. Gadolinium is not required for EFT measurement but for the viability study of the patients.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting for cardiac MRI unit in Assiut University Hospital for viability assessment.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
correlation between EFT volume measured by Cardiac MRI and the angiographic severity of coronary artery disease (Syntax Score) in diabetic vs non diabetic CAD population | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Bakeer Mohamed Bakeer, MSC, Principal Investigator — Assiut University